CLINICAL TRIAL: NCT03169725
Title: A Prospective, Multi-national, Multi-center, Double-blind, Randomized, Active Controlled, Parallel-group, Seamless Phase II/III Clinical Study to Evaluate the Safety and Immunogenicity of 'LBVC (Sabin Poliomyelitis Vaccine (Inactivated))' Compared With 'Imovax® Polio (Poliomyelitis Vaccine (Inactivated))' in Healthy Infants
Brief Title: A Clinical Study to Evaluate the Safety and Immunogenicity of Inactivated Poliomyelitis Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LG-VCCL001
Record Dates: First submitted 2017-05-11; First posted 2017-05-30 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-01

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test group 1 (Experimental): Low dose (Stage2: Lot A) of investigational inactivated poliomyelitis vaccine based on Sabin strains (LBVC)
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strain)
- Test group 2 (Experimental): Middle dose (Stage2: Lot B) of investigational inactivated poliomyelitis vaccine based on Sabin strains (LBVC)
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strain)
- Test group 3 (Experimental): High dose (Stage2: Lot C) of investigational inactivated poliomyelitis vaccine based on Sabin strains (LBVC)
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Sabin strain)
- Comparator (Active Comparator): Cormmercialized inactivated poliomyelitis vaccine based on Sabin strains (Imovax Polio)
  Interventions: Biological: Inactivated Poliomyelitis Vaccine (Salk strain)

INTERVENTIONS:
Biological: Inactivated Poliomyelitis Vaccine (Sabin strain) — Investigational IPV based on Sabin strain (LBVC). Should be injected by intramuscular three injections in the anterolateral aspect of thigh at 6, 10 and 14 weeks of age.
  Arms: Test group 1; Test group 2; Test group 3
Biological: Inactivated Poliomyelitis Vaccine (Salk strain) — Commercialized IPV based on Salk strain (Imovax Polio). Should be injected by intramuscular three injections in the anterolateral aspect of thigh at 6, 10 and 14 weeks of age.
  Arms: Comparator

SUMMARY:
The purpose of the study is to evaluate safety and immunogenicity of inactivated poliomyelitis vaccine based on Sabin strain (LBVC) in healthy infants to select optimal dose of LBVC as well as to demonstrate the lot-to-lot consistency and non-inferiority of LBVC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants of either sex who have reached at least 42 days (6 weeks) of age and not more than 56 days (8 weeks) of age at the time of enrollment
* Born at full term of pregnancy (Gestational age ≥37 weeks)
* Body weight ≥ 3.2 kg at the time of screening
* Born to HIV negative mother
* The parents or Legally Acceptable Representative (LAR) able to understand and comply with planned study procedures
* Signed informed consent by subject's parents or Legally Acceptable Representative (LAR)

Exclusion Criteria:

* Previously received any polio vaccines (OPV or IPV)
* History of previous or concurrent vaccinations other than HepB, BCG, DTP, Hib, Rotavirus vaccine and PCV
* History of bleeding disorder contraindicating intramuscular injection.
* Experienced fever ≥ 38 °C/ 100.4 °F within the past 3 days prior to the screening
* Receipt of immunoglobulin or blood-derived product since birth
* History of allergic reactions to any vaccine components, including excipients and preservatives (neomycin, streptomycin and polymyxin B, etc.)
* Known or suspected immune disorder, or received immunosuppressive therapy
* History of poliomyelitis
* History of any neurological disorders or seizures
* Known or suspected febrile, acute or progressive illness
* Household contact and/or intimate exposure in the previous 30 days to an individual with poliomyelitis
* Participation in another interventional trial within 30 days before to the enrollment or simultaneous participation in another clinical study
* Infants whose families are planning to leave the area of the study site before the end of the study period
* Infants who is considered unsuitable for the clinical study by the investigator

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1417 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Stage1: Seroconversion rate(%) | 4 weeks after 3rd vaccination
  Proportion of subjects achieving seroconversion of each poliovirus serotype using microneutralization assay
Stage2: Seroconversion rate(%) | 4 weeks after 3rd vaccination
  Proportion of subjects achieving seroconversion of each poliovirus serotype using microneutralization assay

SECONDARY OUTCOMES:
Stage1: Seroconversion rate (%) | 4 weeks after 2nd vaccination
  Proportion of subjects achieving seroconversion of each poliovirus serotype using microneutralization assay
Stage2: Seroprotection rate (%) | 4 weeks after 3rd vaccination
  Proportion of subjects achieving seroprotection of each poliovirus serotype using microneutralization assay
Stage1: GMTs (Geometric Mean Titers) | 4 weeks after 2nd and 3rd vaccination
  Comparison of GMTs and GMT ratios
Stage2: GMTs (Geometric Mean Titers) | 4 weeks after 3rd vaccination
  Comparison of GMTs and GMT ratios

CONTACTS AND LOCATIONS:
Locations (3):
- Research Institute for Tropical Medicine, Alabang, Philippines
- Thailand (2):
  - Mahidol University Faculty of Medicine Siriraj Hospital, Bangkok
  - Chiang Mai University Maharaj Nakhon Chiang Mai Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capeding MR, Gomez-Go GD, Oberdorfer P, Borja-Tabora C, Bravo L, Carlos J, Tangsathapornpong A, Uppala R, Laoprasopwattana K, Yang Y, Han S, Wittawatmongkol O. Safety and Immunogenicity of a New Inactivated Polio Vaccine Made From Sabin Strains: A Randomized, Double-Blind, Active-Controlled, Phase 2/3 Seamless Study. J Infect Dis. 2022 Aug 24;226(2):308-318. doi: 10.1093/infdis/jiaa770. PMID 33351072